CLINICAL TRIAL: NCT04383340
Title: Sensitivity Training for Mothers With Premature Infants: A Randomized Controlled Trial
Brief Title: Sensitivity Training for Parents With Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KCC/RC/G/1819-B03
Record Dates: First submitted 2020-05-05; First posted 2020-05-12 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2020-05

CONDITIONS: Premature Birth
Keywords: sensitivity training; mother-infant interaction
MeSH Terms: conditions — Premature Birth | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: All individual assessments were conducted by a clinical psychologist at the hospital who was blinded to the experimental condition of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mother-Infant Transaction Program (Experimental): Four sessions were delivered to the mothers one-on-one based on a manualized protocol while the infants were still in the neonatal intensive care units. These coaching sessions included psychological care for the mother and topics on recognizing premature infant's characteristics, understanding and recognizing signs of infant stress and infant's engagement and disengagement cues, principles of graded stimulation, and how to optimize interactions and avoid over-stimulating the infant.
  Interventions: Behavioral: Mother-Infant Transaction Program
- Treatment as usual (Active Comparator): For this group, infants and mothers received standard hospital care following the initial baseline assessment; these mothers were invited to ask questions about recommended ways to take care of their infants, but no specific knowledge or skills targeted by the adapted MITP program were taught
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Mother-Infant Transaction Program — Parent sensitivity training for mothers of premature infants
  Arms: Mother-Infant Transaction Program
Behavioral: Treatment as usual — Standard hospital care and parental support
  Arms: Treatment as usual

SUMMARY:
This study evaluated the effectiveness of a culturally adapted version of the Mother-Infant Transaction Program (MITP) among Chinese mothers with premature infants in public hospitals in Hong Kong.

DETAILED DESCRIPTION:
Potential participants at two public hospitals in Hong Kong were identified by ward nurses. Mother-infant dyads with infants born at 36 weeks or earlier were assessed for eligibility. Data collection was conducted after obtaining written consent from the mothers. Mother-infant dyads who met the inclusion criteria were randomly allocated to either the intervention or the treatment-as-usual control group. Each dyad was assessed at six time points, i.e., baseline, immediately after intervention/TAU, and when the infants were at the gestation-corrected ages of 3, 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with premature infants born at 36 weeks or earlier

Exclusion Criteria:

* insufficient spoken and written Chinese ability of the mother
* mother under 18 years of age
* triplets or higher multiples
* infants with congenital abnormalities (e.g., metabolic disorder, chromosomal disorder)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Behavioral observation of mother-infant interactions | At baseline prior to intervention
  Maternal sensitivity and quality of mother-infant interaction measured by coding a 5-min video of mother-infant interaction. The coded variables are rated on a 5-point scale, and higher scores indicate higher maternal sensitivity and better interaction quality.
Behavioral observation of mother-infant interactions | Immediately after intervention
  Maternal sensitivity and quality of mother-infant interaction measured by coding a 5-min video of mother-infant interaction. The coded variables are rated on a 5-point scale, and higher scores indicate higher maternal sensitivity and better interaction quality.
Behavioral observation of mother-infant interactions | At infant's corrected age of 3 months
  Maternal sensitivity and quality of mother-infant interaction measured by coding a 5-min video of mother-infant interaction. The coded variables are rated on a 5-point scale, and higher scores indicate higher maternal sensitivity and better interaction quality.
Behavioral observation of mother-infant interactions | At infant's corrected age of 6 months
  Maternal sensitivity and quality of mother-infant interaction measured by coding a 5-min video of mother-infant interaction. The coded variables are rated on a 5-point scale, and higher scores indicate higher maternal sensitivity and better interaction quality.
Maternal postnatal depression | At baseline prior to intervention
  Maternal depression measured by the Edinburgh Postnatal Depression Scale. Possible scores range from 0 to 30. Higher scores indicate higher levels of depression.
Maternal postnatal depression | Immediately after intervention
  Maternal depression measured by the Edinburgh Postnatal Depression Scale. Possible scores range from 0 to 30. Higher scores indicate higher levels of depression.
Maternal postnatal depression | At infant's corrected age of 3 months
  Maternal depression measured by the Edinburgh Postnatal Depression Scale. Possible scores range from 0 to 30. Higher scores indicate higher levels of depression.
Maternal postnatal depression | At infant's corrected age of 6 months
  Maternal depression measured by the Edinburgh Postnatal Depression Scale. Possible scores range from 0 to 30. Higher scores indicate higher levels of depression.
Parenting stress | At baseline prior to intervention
  Parenting stress measured by the Parenting Stress Index-Short Form. Possible scores range from 36 to 180. Higher scores indicate higher levels of parenting stress.
Parenting stress | Immediately after intervention
  Parenting stress measured by the Parenting Stress Index-Short Form. Possible scores range from 36 to 180. Higher scores indicate higher levels of parenting stress.
Parenting stress | At infant's corrected age of 3 months
  Parenting stress measured by the Parenting Stress Index-Short Form. Possible scores range from 36 to 180. Higher scores indicate higher levels of parenting stress.
Parenting stress | At infant's corrected age of 6 months
  Parenting stress measured by the Parenting Stress Index-Short Form. Possible scores range from 36 to 180. Higher scores indicate higher levels of parenting stress.
Infant's temperament | At baseline prior to intervention
  Infant's soothability based on the Infant Behavior Questionnaire. A higher average score denotes higher soothability of the infant, and the highest possible score is 7.
Infant's temperament | Immediately after intervention
  Infant's soothability based on the Infant Behavior Questionnaire. A higher average score denotes higher soothability of the infant, and the highest possible score is 7.
Infant's temperament | At infant's corrected age of 3 months
  Infant's soothability based on the Infant Behavior Questionnaire. A higher average score denotes higher soothability of the infant, and the highest possible score is 7.
Infant's temperament | At infant's corrected age of 6 months
  Infant's soothability based on the Infant Behavior Questionnaire. A higher average score denotes higher soothability of the infant, and the highest possible score is 7.
Infant's weight gain | At infant's corrected age of 3 months
  Infant's weight gain from birth
Infant's weight gain | At infant's corrected age of 6 months
  Infant's weight gain from birth
Infant's weight gain | At infant's corrected age of 9 months
  Infant's weight gain from birth
Infant's weight gain | At infant's corrected age of 12 months
  Infant's weight gain from birth
Infant's developmental outcomes | At infant's corrected age of 3 months
  Measured by the Cognitive Battery of the Merrill-Palmer-Revised Scales of Development, which includes assessments in the cognitive, receptive language, and fine motor domains. Higher scores denote better performance in the assessments
Infant's developmental outcomes | At infant's corrected age of 6 months
  Measured by the Cognitive Battery of the Merrill-Palmer-Revised Scales of Development, which includes assessments in the cognitive, receptive language, and fine motor domains. Higher scores denote better performance in the assessments
Infant's developmental outcomes | At infant's corrected age of 9 months
  Measured by the Cognitive Battery of the Merrill-Palmer-Revised Scales of Development, which includes assessments in the cognitive, receptive language, and fine motor domains. Higher scores denote better performance in the assessments
Infant's developmental outcomes | At infant's corrected age of 12 months
  Measured by the Cognitive Battery of the Merrill-Palmer-Revised Scales of Development, which includes assessments in the cognitive, receptive language, and fine motor domains. Higher scores denote better performance in the assessments

CONTACTS AND LOCATIONS:
Overall Officials: Terry Au, PhD, Study Director — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Derived] Yu NKK, Shum KK, Lam YY, Kwan QKL, Ng SYP, Chan NTT. Sensitivity Training for Mothers With Premature Infants: A Randomized Controlled Trial. J Pediatr Psychol. 2022 Oct 19;47(10):1167-1184. doi: 10.1093/jpepsy/jsac051. PMID 35666133